CLINICAL TRIAL: NCT00789152
Title: The Effects of Desloratadine and Levocetirizine on Nasal Obstruction in Subjects With Induced Allergic Rhinitis in the VCC Assessed Clinically and With Nasal Rhinomanometry and Nasal Flowmetry
Brief Title: The Effect of Desloratadine and Levocetirizine on Nasal Obstruction (Study P03609)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P03609
Record Dates: First submitted 2008-10-30; First posted 2008-11-11 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- desloratadine followed by levocetirizine (Experimental): Subjects in this arm received desloratadine 5 mg daily for 8 days, followed by 10 day washout period, then followed by levocetirizine 5 mg daily for 8 days
  Interventions: Drug: desloratadine; Drug: levocetirizine
- levocetirizine followed by desloratadine (Experimental): Subjects in this arm received levocetirizine 5 mg daily for 8 days, followed by 10 day washout period, then followed by desloratadine 5 mg daily for 8 days
  Interventions: Drug: desloratadine; Drug: levocetirizine

INTERVENTIONS:
Drug: desloratadine — desloratadine 5 mg daily x 8 days
  Other Names: Clarinex, SCH 034117
Drug: levocetirizine — levocetirizine 5 mg daily x 8 days
  Other Names: XYZAL®

SUMMARY:
This was a study to measure the ability of desloratadine and levocetirizine to decrease nasal obstruction in subjects who had study-induced allergic rhinitis. Study participants had allergic rhinitis symptoms induced in a Vienna Challenge Chamber and then received desloratadine or levocetirizine for 8 days. After at least a 10 to 35-day washout period (time when no drug is given), subjects received the opposite treatment for 8 days. Subjects had their total nasal symptom measured.on the 8th day of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Were free of any clinically significant disease that would interfere with study evaluations.
* Demonstrated hypersensitivity to the grass allergen used in the chamber unless confirmed previously within 12 months.
* Hypersensitivity to the allergen was documented by a positive response to the skin prick test with a wheal diameter at least 3 mm larger than the diluent control and by a radioallergosorbent test (RAST) class of >=2 (rating scale 0 -6).
* Had a history of SAR for at least 2 years, as diagnosed by the investigator, another physician, or subject-provided history.
* Reported having shown therapeutic efficacy with previous use of an antihistamine (without a decongestant).
* At the screening allergen provocation, the subject had a nasal obstruction symptom severity score of at least moderate (>=2) and a decrease from baseline in nasal airflow (mL/sec) measured by rhinomanometry of >=30% within 2 hours of allergen exposure. Also, the subject had a nasal obstruction symptom severity score of none or mild (<=1) prior to exposure to allergen.

Exclusion Criteria:

* Women who were pregnant or nursing.
* Had a body mass index (BMI) >=30 kg/m^2.
* Had asthma; were being treated with inhaled or oral corticosteroids, chromones, theophylline, leukotriene inhibitors, or short-acting inhaled β2-agonists (except during or immediately after the allergen exposures); and could not go through the washout periods and the entire study without needing these medications.
* Developed wheezing or dyspnea during the screening allergen exposure.
* Had a respiratory infection during the 4 weeks prior to pre-dose evaluations.
* Had any clinically significant deviation from normal in the physical examination that, in the investigator's judgment, could interfere with the study evaluation or affect subject safety.
* Had any history of or laboratory evidence of hepatic failure or renal failure with a glomerular filtration rate (GFR) known to be <30 mL/min.
* Had a known potential for hypersensitivity, allergic, or idiosyncratic reaction to the study drug or excipients.
* Had nasal structural abnormalities, including large nasal polyps and marked septum deviation, that significantly interfered with nasal airflow.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2003-12-01 (Actual); Primary Completion 2004-05-01 (Actual); Study Completion 2004-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score (TNSS) at the end of treatment phase compared to pre-exposure baseline scores | End of each treatment phase (8th day)

SECONDARY OUTCOMES:
Nasal Peak Inspiratory Flow (NPIF), Nasal secretion weights, nasal airflow, individual nasal symptoms, TNSS, Total Non-Nasal Symptoms Severity Score (TNNSS), Total Symptom Score (TSS) | End of each treatment phase (8th day)
Safety | All study visits